CLINICAL TRIAL: NCT06655467
Title: Understanding Psychological Distress and Therapeutic Environment in the Emergency Department
Acronym: UPDATE-ED
Status: Not yet recruiting | Type: Observational
Sponsor: NHS Fife (Other Government)
Collaborators: Royal College of Emergency Medicine (Other)
Responsible Party: Principal Investigator, Rajendra Raman, Chief Investigator, NHS Fife
Other Study IDs: 24/EM/0245
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Mental Health; Substance Use (Drugs, Alcohol); Psychological Distress
MeSH Terms: conditions — Psychological Well-Being; Substance-Related Disorders | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: Routine Care — This study involves no change in clinical care and no study specific interventions for participants.
  Other Names: Standard Care

SUMMARY:
This research aims to establish the number of patients coming to Emergency Departments (EDs) with issues relating to mental health, alcohol or drugs, or in some form of psychological distress, including those for whom this was not the main reason for attending ED. We will collect anonymous information on age, gender, ethnicity, when and how they came to the ED, where and how they are cared for whilst in the ED, and what happens to them afterwards. With this information we hope to build a better picture of these patients so we can go on to design and test ways to improve their care in the future.

DETAILED DESCRIPTION:
Those presenting to the Emergency Department with mental ill health, substance misuse or in crisis have a worse patient journey than those presenting with physical issues alone. They wait twice as long to be seen1 and have poorer experiences. Recognising this, the RCEM/James Lind Alliance Priority Setting Partnership has placed mental health at the top of the Emergency Medicine research agenda. The question asked is: "How can care for mental health patients be optimised, whether presenting with either/both physical and mental health needs; including appropriate space to see patients, staff training, early recognition of symptoms, prioritisation, and patient experience?" An explicit research agenda has yet to emerge from this very broad question. At the most basic level, the patient population needs to be defined, the scale of the problem quantified, and current practice patterns and variation described in detail.

It has been estimated that the proportion of ED attendances related to "mental health disorders" is 4%. However these estimates are derived from retrospective data and are dependent on accurate diagnosis coding. There is a lack of data on dual diagnoses, which Scotland's Mental Health strategy has outlined as a key area for action, recommending opportunities to "pilot improved arrangements for dual diagnosis for people with problem substance use and mental health diagnosis". A literature review aiming to build a 'Typology' of psychiatric emergency services in the UK emphasised wide variation in provision and heterogeneity of models. No prospective study has yet quantified this variation in terms of waiting times, types of assessment offered, disposition and outcomes. The success of other large observational studies on ED presentations such as syncope, acute aortic syndromes and frailty suggests that a similar methodology could be applied to mental health and related presentations.

ELIGIBILITY:
Inclusion Criteria:

* Issues of mental health AND/OR
* Issues of substance use AND/OR
* Psychological distress (this refers to patients without an established mental health or substance use disorder who nonetheless present in a distressed state, where distress is not caused by a readily identifiable and treatable physical condition) AND/OR
* Where the treating ED team feel the patient would benefit from some form of mental health or addictions assessment or intervention, whether carried out by ED staff, specialist services or third sector agencies.

Exclusion Criteria:

1. Patients aged 10 and under.
2. Patients with distress caused by a physical condition, relieved by appropriate treatment.
3. Delirium, unless caused by a mental health- or substance-related disorder.
4. Patients with alcohol intoxication alone, without other evidence of harmful use of alcohol and without evidence of psychological distress.

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting to the Emergency Department (ED) with issues of mental health, substance use or psychological distress, whether or not this was the primary reason for presentation.
Sampling Method: Non-Probability Sample
Enrollment: 398 (Estimated)
Dates: Start 2025-02-03 (Estimated); Primary Completion 2025-03-18 (Estimated); Study Completion 2025-03-18 (Estimated)

PRIMARY OUTCOMES:
Proportion fo ED attendance related to issues of mental health, substance use or psychological distress | 7 days
  Number of patients meeting eligibility criteria, expressed as a proportion of all ED attendances at each site during the study period.

SECONDARY OUTCOMES:
Proportion of patients physically in ED who meet inclusion criteria at any one time | 7 days
  Proportion of patients physically in the ED who meet inclusion criteria at any given time over the 7-day study period.
Comparison with coding data | 7 days
  Proportion of total ED patients meeting inclusion criteria during the study period compared with coding data from a recent historical cohort at one site (NHS Fife).
Admission rate | 7 days
  Proportion of patients meeting inclusion criteria who are admitted to hospital on an informal basis, and proportion admitted under detention.
Length of stay | 30 days
  Mean, standard deviation (or nonparametric equivalents) and range of lengths of ED and hospital stay for patients meeting inclusion criteria.
Specialist mental health or addictions input in ED | 7 days
  Proportion of patients meeting inclusion criteria who receive specialist mental health or addictions input whilst in ED.
Specialist referrals from ED | 7 days
  Proportion of patients meeting inclusion criteria who are referred by the ED team for specialist mental health or addictions input after ED discharge.
7-day and 30-day follow-up | 30 days
  Proportion of patients meeting inclusion criteria who return to ED, are admitted to hospital or die within 7 and 30 days of index ED visit.
Clinician Confidence Scale | 7 days
  Self-reported confidence of ED clinicians (Visual Analog Scale) in managing an individual patient presenting with issues of mental health, substance use or psychological distress. Values may range from 0 (no confidence at all) to 10 (complete confidence).
Resource Availability Scale | 7 days
  Perception of resource availability (self-reported by ED clinicians on a Visual Analog Scale) for managing an individual patient presenting with issues of mental health, substance use or psychological distress. Values may range from 0 (complete lack of resources) to 10 (all resources available).

CONTACTS AND LOCATIONS:
Locations (1):
- Victoria Hospital, Kirkcaldy, Fife, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Background] European Taskforce on Geriatric Emergency Medicine (ETGEM) collaborators. Prevalence of Frailty in European Emergency Departments (FEED): an international flash mob study. Eur Geriatr Med. 2024 Apr;15(2):463-470. doi: 10.1007/s41999-023-00926-3. Epub 2024 Feb 10. PMID 38340282
- [Background] McLatchie R, Reed MJ, Freeman N, Parker RA, Wilson S, Goodacre S, Cowan A, Boyle J, Clarke B, Clarke E; DAShED investigators. Diagnosis of Acute Aortic Syndrome in the Emergency Department (DAShED) study: an observational cohort study of people attending the emergency department with symptoms consistent with acute aortic syndrome. Emerg Med J. 2024 Feb 20;41(3):136-144. doi: 10.1136/emermed-2023-213266. PMID 37945311
- [Background] Reed MJ, Karuranga S, Kearns D, Alawiye S, Clarke B, Mockel M, Karamercan M, Janssens K, Riesgo LG, Torrecilla FM, Golea A, Fernandez Cejas JA, Lupan-Muresan EM, Zaimi E, Nuernberger A, Rennet O, Skjaerbaek C, Polyzogopoulou E, Imecz J, Groff P, Camilleri R, Cimpoesu D, Jovic M, Miro O, Anderson R, Laribi S; SEED investigators. Management of syncope in the Emergency Department: a European prospective cohort study (SEED). Eur J Emerg Med. 2024 Apr 1;31(2):136-146. doi: 10.1097/MEJ.0000000000001101. Epub 2023 Nov 27. PMID 38015745
- [Background] Odejimi O, Bagchi D, Tadros G. Typology of psychiatric emergency services in the United Kingdom: a narrative literature review. BMC Psychiatry. 2020 Dec 10;20(1):587. doi: 10.1186/s12888-020-02983-5. PMID 33302905
- [Background] Scottish Government (2017) Mental Health Strategy: 2017-2027. Crown Copyright. Available at: https://www.gov.scot/binaries/content/documents/govscot/publications/strategy-plan/2017/03/mental-health-strategy-2017-2027/documents/00516047-pdf/00516047-pdf/govscot%3Adocument/00516047.pdf
- [Background] Barratt H, Rojas-Garcia A, Clarke K, Moore A, Whittington C, Stockton S, Thomas J, Pilling S, Raine R. Epidemiology of Mental Health Attendances at Emergency Departments: Systematic Review and Meta-Analysis. PLoS One. 2016 Apr 27;11(4):e0154449. doi: 10.1371/journal.pone.0154449. eCollection 2016. PMID 27120350
- [Background] Baracaia S, McNulty D, Baldwin S, Mytton J, Evison F, Raine R, Giacco D, Hutchings A, Barratt H. Mental health in hospital emergency departments: cross-sectional analysis of attendances in England 2013/2014. Emerg Med J. 2020 Dec;37(12):744-751. doi: 10.1136/emermed-2019-209105. Epub 2020 Nov 5. PMID 33154100
- [Background] Royal College of Emergency Medicine (2022) James Lind Alliance Emergency Medicine Priority Setting Partnership Refresh 2022. Available at: https://rcem.ac.uk/research-priorities/
- [Background] Digel Vandyk A, Young L, MacPhee C, Gillis K. Exploring the Experiences of Persons Who Frequently Visit the Emergency Department for Mental Health-Related Reasons. Qual Health Res. 2018 Mar;28(4):587-599. doi: 10.1177/1049732317746382. Epub 2017 Dec 12. PMID 29231128
- [Background] Clarke DE, Dusome D, Hughes L. Emergency department from the mental health client's perspective. Int J Ment Health Nurs. 2007 Apr;16(2):126-31. doi: 10.1111/j.1447-0349.2007.00455.x. PMID 17348963
- [Background] Royal College of Emergency Medicine (2022) RCEM Acute Insight Series: Mental Health Emergency Care. Available at: https://rcem.ac.uk/wp-content/uploads/2022/09/RCEM-Acute-Insight-Series-Mental-Health-Emergency-Care.pdf